CLINICAL TRIAL: NCT00068068
Title: Safety and Efficacy of Treating Refractory Cancers With the Litx™ System: Phase II Safety and Efficacy Study in Patients With Liver Metastases From Colorectal Cancer That Have Failed Chemotherapy
Brief Title: Photodynamic Therapy With Talaporfin Sodium (LS11) in Treating Patients With Refractory Colorectal Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Light Sciences LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSC-OL002; NCT00078871 (obsolete NCT alias)
Record Dates: First submitted 2003-09-04; First posted 2003-09-08 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Liver Metastasis; Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis
Keywords: Photodynamic therapy; Liver metastases; Colorectal cancer; Litx™; Light Infusion Technology™; Talaporfin sodium; LS11; Liver mets; Metastatic colorectal cancer; Light emittting diodes (LED); Tumor ablation; Combination therapy
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis | interventions — Talaporfin; Photochemotherapy; Phototherapy; Drug Therapy

INTERVENTIONS:
Drug: Talaporfin sodium (LS11)
Device: LED-based light infusion device
Device: Light emitting diodes (LED)
Procedure: Photodynamic therapy
Procedure: Phototherapy
Procedure: Chemotherapy

SUMMARY:
The purpose of this study is to determine whether the Litx platform is safe and effective in the treatment of liver metastasis arising from colorectal cancer. Litx is a next-generation photodynamic therapy platform in which the drug, talaporfin sodium (LS11), is activated by light from the light-emitting diode (LED)-based light infusion device, inserted directly into the tumor through the skin prior to treatment.

DETAILED DESCRIPTION:
Patients that provide Informed Consent and satisfy the Eligibility Criteria will undergo CT or ultrasound guided percutaneous placement of a single, two, three, or four light infusion devices depending on their tumor characteristics. No more than 4 light sources will be used at a single treatment. The light infusion devices may be used in a single lesion or in multiple lesions.

Following radiographic confirmation of light infusion device placement, patients will receive an intravenous dose of LS11 at 40 mg/m². One hour following completion of LS11 administration, delivery of 200 J/cm light energy will begin. The light infusion device will then be manually removed and the patients will be observed for acute complication of light infusion device removal. Precautions for protection from external light exposure should be instituted beginning with the LS11 administration and be maintained as defined throughout the study period. On day 30+5 the patient will undergo clinical assessment and the tumor mass will be imaged using contrast enhanced spiral CT for determination of volume and radius of the tumor size, as well as tumor necrosis. The patient may then receive 5-FU and/or leucovorin + either irinotecan or oxaliplatin standard chemotherapy at day 30 visit. All patients, with or without chemotherapy at day 30, will undergo final clinical assessment and final tumor imaging evaluation using contrast CT at day 60+5 of Litx treatment.

ELIGIBILITY:
Inclusion Criteria

* Patients with metastatic liver lesions from colorectal disease who have failed or progressed on a chemotherapy regimen for metastatic disease.
* Biopsy proven evidence of colorectal cancer.
* Patients with 4 or fewer lesions greater than 1 cm and with no single lesion greater than 7 cm in maximum diameter.
* Age greater than or equal to 18 years.
* Patients must be able to sign informed consent.
* Life expectancy greater than or equal to 3 months.
* ECOG performance status 0-2.
* Patients with extrahepatic disease in addition to their hepatic metastases are eligible and will receive systemic therapy for their extrahepatic disease following Litx therapy.
* Off chemotherapy for 4 weeks. Must have recovered from the chemotherapy effects.

Exclusion Criteria

Patients must be excluded if any of the following apply:

* Patients who are candidates for complete surgical resection.
* Pregnancy or breast-feeding. A negative pregnancy test (urine or serum) is required prior to enrollment.
* Known uncontrollable serious reactions such as anaphylaxis, to the contrast agents used in this study.
* PT or PTT greater than 1.5X control.
* Platelet count less than 100,000.
* WBC less than 2500/mm.
* Neutrophils less than 2000/mm.
* Hemoglobin less than 9 g/dL.
* Liver enzymes greater than 3 X ULN.
* Total bilirubin greater than 1.5 X ULN.
* Serum creatinine greater than 2.5 X ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - HealthOne Alliance/Presbyterian St. Lukes Medical Center, Denver, Colorado
  - Eastern Carolina University, School of Medicine, Greenville, North Carolina
  - University of Pennsylvania / Department of Radiation Oncology, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
- University Hospital Frankfurt, Johann Wolfgang Goethe-University, Frankfurt am Main, Germany

REFERENCES:
- [Background] Chen J, Keltner L, Christophersen J, Zheng F, Krouse M, Singhal A, Wang SS. New technology for deep light distribution in tissue for phototherapy. Cancer J. 2002 Mar-Apr;8(2):154-63. doi: 10.1097/00130404-200203000-00009. PMID 11999949
- [Background] Lustig RA, Vogl TJ, Fromm D, Cuenca R, Alex Hsi R, D'Cruz AK, Krajina Z, Turic M, Singhal A, Chen JC. A multicenter Phase I safety study of intratumoral photoactivation of talaporfin sodium in patients with refractory solid tumors. Cancer. 2003 Oct 15;98(8):1767-71. doi: 10.1002/cncr.11708. PMID 14534895
- See also: Sponsor website — http://www.lightsciences.com